CLINICAL TRIAL: NCT06518746
Title: Gonadal Dysgenesis Tissue Cryopreservation for Fertility Preservation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-3159
Record Dates: First submitted 2024-07-03; First posted 2024-07-24 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryopreservation of gonadal tissue (Experimental): Enrolled participants will undergo gonadal tissue processing, freezing and cryopreservation after the standard care (gonadectomy, gonadal tissue histologic examination)
  Interventions: Other: Cryopreservation of gonadal tissue

INTERVENTIONS:
Other: Cryopreservation of gonadal tissue — Patients at risk for primary gonadal tumors will undergo unilateral or bilateral gonadectomy for clinical purposes as a standard of care, and a portion of the surgically removed tissue will be cryopreserved for fertility preservation. The pathologist will assess the tissue using sterile technique and every other section will undergo histologic analysis, including evaluation for the presence of tumor or viable germ cell elements. The sections of the tissue for fertility preservation will be refrigerated and held until a final diagnosis is made on the tissue sections that are being processed for histologic analysis. If no tumor is identified and viable germ cell elements are identified, the tissue sections allotted for preservation will be sent in holding media for processing and cryopreservation.

SUMMARY:
The "Gonadal Dysgenesis Tissue Cryopreservation for Fertility Preservation" study is open to a subset of patients with disorders of sex development (DSD) which is associated with the risk of malignancy and a high risk of infertility or sterility. For these patients, experimental gonadal tissue cryopreservation is the only fertility preservation option available. The overall objective of this study is to determine the safety and efficacy of gonadal tissue cryopreservation as a method of preserving fertility and/or restoring hormonal function in patients with gonadal dysgenesis who are at risk of decreased fertility potential or malignancy.

DETAILED DESCRIPTION:
Unlike the oncology population, in which patients have inherently normal fertility potential and reproductive function, individuals with DSD may have infertility caused by 1) abnormal gonadal development, 2) gonadectomy performed for risk of malignancy, 3) abnormal hormone production or, 4) discordance, or difference, between gonadal type and gender identity. Fertility potential differs according to the specific DSD diagnosis and can also be influenced by age, genetic mosaicism, and/or risk of developing a gonadal malignancy.

Abnormal gonadal development can result in gonadal failure, either in infancy or progressively, such that individuals may not undergo spontaneous puberty, menarche or spermarche. Progressive germ cell loss may occur throughout childhood. In addition, abnormal gonadal development in certain cellular environments leads to an increased risk of germ cell cancer. Traditionally, it was recommended to perform gonadectomy at the time of diagnosis in all DSD conditions with a risk of gonadal tumor formation. The estimated tumor risk ranges from 2% in complete androgen insensitivity syndrome to 40% in partial androgen insensitivity syndrome. Advances in stratification of tumor risk have led to a more diagnosis-specific assessment of risk, but tumor risk remains a major concern.

Thus, the investigators are conducting a pilot study to assess the safety and efficacy of gonadal tissue cryopreservation as a method of preserving fertility and/or restoring hormonal function in patients with gonadal dysgenesis who are at risk of decreased fertility potential or malignancy.

ELIGIBILITY:
Inclusion Criteria:

* < 30 years of age
* Individuals diagnosed with a disorder of sex development who have any risk for malignancy in their gonadal tissue and will have their gonads removed for a clinical indication
* Individuals diagnosed with a disorder of sex development who are at risk of primary ovarian insufficiency (POI) due to an underlying genetic condition

Exclusion Criteria:

* Pregnancy
* Patients likely to retain inherent fertility and reproductive function
* Patients deemed high risk for perioperative complications
* Patients 7-17 years of age unable to provide assent (i.e. significant psychiatric problems/cognitive delay)
* Patients 18 and older unable to provide consent (i.e. significant psychiatric problems/cognitive delay)

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy, as Assessed via the Proportion of total samples containing viable gonadal tissue and/or the presence of germ cells, and the Proportion of total samples that were successfully cryopreserved for the patient's future use. | Up to 48 hours after obtaining gonadal tissue samples.
  Determine the efficacy of gonadal tissue and germ cells cryopreservation for patients' future use to restore fertility and/or hormone function. Efficacy is defined as at least 30% of patients having viable gonadal tissue and/or germ cells present.
Safety, as Assessed via the Proportion of adverse events | within 72 hours of gonadal tissue removal
  Number and proportion of adverse events in gonadal tissue cryopreservation
Acceptability as a fertility preservation method, as Assessed via the survey responses by eligible patients and/or their guardians. | Through study completion, up to ten years.
  Descriptive analysis of survey responses, including the Decision Regret Scale scores (mean/median scores across domains).
Level of demand | Through study completion, up to ten years.
  Descriptive analysis of the proportion of eligible patients who elect gonadal tissue cryopreservation (numerator) out of those who are eligible (denominator).

SECONDARY OUTCOMES:
Create a recruitment database of patients/caregivers that consent to future contact to consider participating in other research studies pertaining to fertility preservation. | Through study completion, up to ten years.
  Descriptive analysis of the proportion of patients providing additional consent for future
Determine if there are disparities in the type of patients consenting to future contact for research studies pertaining to fertility preservation | Through study completion, up to ten years.
  Descriptive analysis of the type of patients (including but not limited to age, race, ethnicity, insurance type, medical history/diagnosis) who elect to be contacted for future research opportunities. A Pearson Chi-squared test can be used to examine if this proportion varies across groups. A 2-sample t-test can be used to compare age (continuous) between those who consent to future research and those who did not.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Corkum, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No